CLINICAL TRIAL: NCT00302757
Title: Multicenter Phase I/II Study of Radioimmunotherapy With 90Y-ibritumomab Tiuxetan in a Nonmyeloablative Conditioning Regimen for Allogeneic Hematopoietic Cell Transplantation From HLA-identical Donors in Patients With Advanced Non-Hodgkin Lymphoma
Brief Title: Radioimmunotherapy With 90Y-ibritumomab Tiuxetan as Part of a Dose Reduced Conditioning Regimen for Allogeneic Hematopoietic Cell Transplantation for the Treatment of Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002206-37
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: NHL; low and high grade non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Radioimmunotherapy

INTERVENTIONS:
Drug: Radioimmunotherapy
Procedure: allogeneic hematopoietic cell transplantation

SUMMARY:
The study evaluates the additional use of radioimmunotherapy with a 90-Yttrium labeled monoclonal antibody targeting lymphoma cells in two dose reduced conditioning regimens for allogeneic hematopoietic cell transplantation from human leukocyte antigen (HLA)-identical donors. Radioimmunotherapy should allow an increased anti-lymphoma effect of the conditioning while the allogeneic grafts may confer potent graft versus lymphoma effects and rescue from potential hematopoietic side effects of the radioimmunotherapy. The study evaluates the feasibility and toxicity of such approach and will also analyze disease response and survival of the patients treated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced CD20+ NHL (non-Hodgkin lymphoma) relapsed after at least two preceding chemotherapy regimens including treatment with rituximab or with relapse after autologous HCT (hematopoietic cell transplantation)

The following entities of lymphomas can be included in Arm A of the protocol:

Arm A:

* Small lymphocytic lymphoma (SLL/CLL)
* Mantle cell lymphoma (MCL)
* Follicular lymphoma Grade 1-2
* Marginal zone lymphoma (MZL)

  * Extranodal (MALT lymphoma)
  * Nodal (Monocytoid B-cell lymphoma)
  * Splenic

The following lymphoma entities can be included in Arm B of the protocol:

Arm B:

* Diffuse large B-cell lymphoma/follicular lymphoma grade 3
* Grade 3 follicular lymphoma
* Blastic mantle cell lymphoma
* Mediastinal B-cell lymphoma

  * Age > 18, < 70 years
  * Karnofsky score > 60%
  * HLA-identical related or unrelated donor
  * CD20+ lymphoma cells on biopsy or peripheral blood
  * Disease stage at inclusion: CR, PR or SD

Exclusion Criteria:

* Patients with rapidly progressive disease
* Less than 3 months after preceding HCT
* CNS involvement with disease
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Liver function abnormalities with bilirubin > 2 mg/dL and elevation of transaminases higher than 2x upper limit of normal
* Chronic active viral hepatitis
* Ejection fraction < 40% on echocardiography
* Patients with > grade II hypertension by CTC criteria
* Creatinine clearance < 50 ml/min
* Respiratory failure necessitating supplemental oxygen or DLCO < 30%
* Allergy against murine antibodies
* HIV infection
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control during study treatment and for at least 12 months thereafter. (Women of childbearing potential must have a negative serum pregnancy test at study entry.)
* Patients with pleural effusion or ascites
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Patients who received any investigational drugs less than 4 weeks before entry in this study or who have not as yet recovered from the toxic effects of such therapy
* Patients who underwent surgery within 4 weeks of entering the study or patients who have not as yet recovered from the side-effects of such treatment
* Patients with a history of psychiatric illness or condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol
* Unable to give informed consent
* Enrollment in another trial interfering with the endpoints of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
treatment related toxicity
engraftment

SECONDARY OUTCOMES:
disease response
relapse rate
disease free survival
overall survival
graft versus host disease (GVHD)
immunoreconstitution

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A Bethge, MD, Principal Investigator — Medical Center University of Tuebingen; Donald Bunjes, MD, Principal Investigator — Medical Center University of Ulm
Locations (11):
- Germany (11):
  - Medical Center Charite Benjamin Franklin, Berlin
  - University of Dresden Medical Center, Dresden
  - Center for Marrow Transplantation, University of Essen, Essen
  - Medical Center University of Goettingen, Göttingen
  - Medical Center University of Hannover, Hanover
  - Medical Center University of Leipzig, Leipzig
  - Medical Center University of Muenster, Münster
  - South West German Cancer Center, University of Tuebingen Medical Center, Tübingen
  - Medical Center University of Ulm, Ulm
  - Stiftung Deutsche Klinik für Diagnostik GmbH, Wiesbaden
  - University of Wuerzburg Medical Center, Würzburg

REFERENCES:
- [Derived] Bethge WA, von Harsdorf S, Bornhauser M, Federmann B, Stelljes M, Trenschel R, Baurmann H, Dittmann H, Faul C, Vogel W, Kanz L, Bunjes D. Dose-escalated radioimmunotherapy as part of reduced intensity conditioning for allogeneic transplantation in patients with advanced high-grade non-Hodgkin lymphoma. Bone Marrow Transplant. 2012 Nov;47(11):1397-402. doi: 10.1038/bmt.2012.62. Epub 2012 Apr 16. PMID 22504934
- [Derived] Bethge WA, Lange T, Meisner C, von Harsdorf S, Bornhaeuser M, Federmann B, Stadler M, Uharek L, Stelljes M, Knop S, Wulf G, Trenschel R, Vucinic V, Dittmann H, Faul C, Vogel W, Kanz L, Bunjes D. Radioimmunotherapy with yttrium-90-ibritumomab tiuxetan as part of a reduced- intensity conditioning regimen for allogeneic hematopoietic cell transplantation in patients with advanced non-Hodgkin lymphoma: results of a phase 2 study. Blood. 2010 Sep 9;116(10):1795-802. doi: 10.1182/blood-2010-02-270538. Epub 2010 Jun 7. PMID 20530284
- See also: Related Info — http://www.onkologie-tuebingen.de